CLINICAL TRIAL: NCT03207880
Title: Piloting an Innovation to Improve the Quality of Remote Abortion Services: Incorporating Use of Multi-Level Pregnancy Tests
Brief Title: Piloting Use of Multi-Level Pregnancy Tests in Remote Abortion Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: safe2choose (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6011
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Medical Abortion, Complete or Unspecified, Without Complication
Keywords: pregnancy test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MLPT (Experimental): Multi-level pregnancy test
  Interventions: Device: Multi-level pregnancy test

INTERVENTIONS:
Device: Multi-level pregnancy test — Study participants will be instructed to perform a baseline MLPT immediately prior to administering the first dose of abortion medication and a second MLPT one week later to ascertain the follow-up hCG range. Any woman who obtains a stable or increasing hCG result, when comparing the baseline test result with the follow-up test result, will be instructed to contact safe2choose. Any woman who obtains a decrease in her hCG range, when comparing the baseline test result with the follow-up test result, will be informed that her abortion was a success and she is no longer pregnant.

SUMMARY:
Serial use of urine multi-level pregnancy tests (MLPTs) has been shown to be a reliable and efficient strategy for excluding ongoing pregnancy after medical abortion at ≤ 63 days of gestation. This pilot project will assess whether MLPTs can enhance the quality of remote medical abortion services through enabling women to reliably ascertain their abortion outcomes at home sooner than would otherwise have been the case.

safe2choose provides remote medical abortion services through the Internet (information, counselling and access to abortion pills) in a growing number of countries worldwide. safe2choose will collaborate with Gynuity Health Projects to pilot the utility of MLPTs for home follow-up as part of its remote medical abortion services.

As safe2choose does not have a physical office, the location of the sponsor's office is listed in this entry as the study location. Women from the United States are NOT eligible to enroll.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of safe2choose medical abortion services
* Able to read English or Spanish
* ≤ 56 days LMP
* Willing and able to read and sign consent form
* Agree to comply with the study procedures, including completing the follow-up survey

Exclusion Criteria:

* Does not meet inclusion criteria

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Proportion of women who successfully receive the MLPTs | 1 week after mailing the MLPTs
Proportion of women who use the MLPTs to determine their abortion outcome | 2 weeks after receiving medical abortion package
Proportion of women able to use MLPTs on their own without guidance or instruction from providers | 2 weeks after receiving medical abortion package
Proportion of women who take action based on the interpretation of their test results | 2 weeks after receiving medical abortion package
Proportion of women who are satisfied with using MLPTs | 2 weeks after receiving medical abortion package

SECONDARY OUTCOMES:
Proportion of all eligible safe2choose clients who elect to participate in the study | 0 days after recruitment
Proportion of women who find the MLPT instructions (written and video) to be helpful tools | 2 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Erica Chong, MPH, Principal Investigator — Gynuity Health Projects; Jennifer Blum, MPH, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Gynuity Health Projects, New York, New York, United States